CLINICAL TRIAL: NCT02925637
Title: Effectiveness of a Novel Meta-cognitive-functional Intervention (FACoT) for Individuals Post Mild-moderate Stroke
Brief Title: Effectiveness of FACoT for Individuals Post Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bait Balev Hospital (Other)
Collaborators: Tel Aviv University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: adamit_t
Record Dates: First submitted 2016-08-03; First posted 2016-10-06 (Estimated); Last update posted 2021-04-14 (Actual); Status verified 2019-02

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FACoT group (Experimental): treatment group will receive FACoT, that include one to one 10 treatment sessions. the treatment sessions will include: functional activities, cognitive activities and strategies (pencil-pen treatment), and behavioural strategies
  Interventions: Other: FaCoT
- control group (No Intervention): control group receiving standard care - cognitive and functional assesment

INTERVENTIONS:
Other: FaCoT — The intervention will include: functional activities, cognitive activities and strategies (pencil-pen treatment), and behavioural strategies
  Arms: FACoT group

SUMMARY:
To develop and assess the effectiveness of a novel cognitive-functional intervention (FACoT) in occupational therapy for people after mild to moderate stroke.

ELIGIBILITY:
inclusion criteria:

* >18 years
* at least three years post stroke
* severity mild to moderate (NIHSS≤5)
* independent prior to the stroke
* can understand and speak Hebrew

Exclusion Criteria:

* with no other neurological or psychiatric conditions
* without dementia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2017-03-12 (Actual); Primary Completion 2020-02-27 (Actual); Study Completion 2020-02-27 (Actual)

PRIMARY OUTCOMES:
Change in scores of The Canadian Occupational Performance Measure (COPM) | Change between baseline (week 0) to time 1 (post-intervention -10-13 weeks later) and time 2 (follow-up- three month later)

SECONDARY OUTCOMES:
Change in scores of the Instrumental Activities of Daily Living (IADL) scale | Change between baseline (week 0) to time 1 (post-intervention, 10-13 weeks later) and between baseline to time 2 (follow-up- 3 month later)
Change in scores of Reintegration to Normal Living Index (RNL) | Change between baseline (week 0) to time 1 (post-intervention, 10-13 weeks later) and between baseline to time 2 (follow-up-3 month later)
Change in scores of Short Form-12v2 Health Survey (SF-12v2) | Change between baseline (week 0) to time 1 (post-intervention, 10-13 weeks later) and between baseline to time 2 (follow-up- 3 month later)
change in scoe of New general self efficacy scale (NGSE) | Change between baseline (week 0) to time 1 (post-intervention, 10-13 weeks later) and between baseline to time 2 (follow-up- 3 month later)
Change in scores of Patient competency rating scale (PCRS) | Change between baseline (week 0) to time 1 (post-intervention, 10-13 weeks later) and between baseline to time 2 (follow-up- 3 month later)
Change in scores Self Regulation Skills Interview (SRSI) | Change between baseline (week 0) to time 1 (post-intervention, 10-13 weeks later) and between baseline to time 2 (follow-up- 3 month later)
Change in scores of Montreal Cognitive Assessment (MoCA) | Change between baseline (week 0) to time 1 (post-intervention, 10-13 weeks later) and between baseline to time 2 (follow-up-3 month later)
Change in scores of Trail making test (TMT) | Change between baseline (week 0) to time 1 (post-intervention, 10-13 weeks later) and between baseline to time 2 (follow-up- 3 month later)
Change in scores of zoo-map | Change between baseline (week 0) to time 1 (post-intervention, 10-13 weeks later) and between baseline to time 2 (follow-up-3 month later)
Change in scores of Dysexecutive Questionnaire (DEX) | Change between baseline (week 0) to time 1 (post-intervention, 10-13 weeks later) and between baseline to time 2 (follow-up- 3month later)
Geriatric Depression Scale - short form (GDS-SF) | Change between baseline (week 0) to time 1 (post-intervention, 10-13 weeks later) and between baseline to time 2 (follow-up- 3 month later)

OTHER OUTCOMES:
National Institutes of Health Stroke Scale (NIHSS) | baseline (week 0)
Functional Independence Measure (FIM) | baseline (week 0)
demographic questionnaire | baseline (week 0)

CONTACTS AND LOCATIONS:
Overall Officials: tal adamit, PHD student, Principal Investigator — Maccabbi health center ashdod isreal
Locations (1):
- Maccabi, Ashdod, Israel

IPD SHARING:
Plan to Share IPD: No